CLINICAL TRIAL: NCT02921425
Title: Use of the Track Health Function of the MyHealtheVet Personal Health Record
Brief Title: Use of Track Health Function of the MyHealthevet Personal Health Record
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 13-135
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Prediabetic State
Keywords: lifestyle; patient health record; Veterans; prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Health Records, Personal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patient health record (Experimental): The study intervention involved the provision to study participants of targeted instruction and practice on use of the Track Health function of the VA's patient health record known as My HealthyVet.
  Interventions: Behavioral: patient health record

INTERVENTIONS:
Behavioral: patient health record — The study intervention involved the provision to study participants of targeted instruction and practice on use of two features of the Track Health (TH) function of the VA's patient health record (PHR) known as My HealthyVet (MHV) -- Journals and Vitals + Readings -- as a basis for promoting positive physical activity (PA) and dietary lifestyles. Seven interactive multimedia instructional modules were developed by the study team. These modules demonstrated on a computer screen how to enter PA and diet information into the Journals feature; how to add weight data into the Vitals + Readings feature; how to view these and other measures in tabular and graphical formats over different time frames; and the concept of possible cause-effect links between behavioral lifestyle and physiological outcome data. Participants were directed to enter food intake, PA, and weight information a specified number of times per week over the 3-month study period.

SUMMARY:
This study was a pilot 3-month clinical trial that investigated the feasibility, effectiveness, and acceptability of using the Track Health function of the Veterans Health Administration's patient health record for effecting a more positive physical activity (PA) and dietary intake lifestyle in a sample of 38 overweight and obese Veterans with prediabetes. Baseline and three-month post-intervention outcomes were measured in two main domains: objective (e.g., weight) and subjective (e.g., self-efficacy).

DETAILED DESCRIPTION:
This was a pilot clinical trial that used a single-group design to test the feasibility, effectiveness, and acceptability of using the Track Health (TH) function of My HealtheVet, the VA's patient health record (PHR), as a tool for effecting a more positive physical activity (PA) and dietary intake lifestyle in overweight and obese Veterans with prediabetes. Baseline and three-month post-intervention outcomes were measured in two main domains: objective (PA as measured by an accelerometer, diet, weight, abdominal circumference, BMI, and blood pressure) and subjective (self-efficacy, intent to adhere to lifestyle change, and patient activation). Assessments, including screening on inclusion and exclusion criteria, physiological measurements, administration of questionnaires, and training on use of two critical features of the TH function--the use of Journals to enter dietary and PA data and the use of Vitals + Readings to enter weight and track physiological measures--took place place across four visits to the study site, which was the Veterans Administration Medical Center in Miami. The investigators hypothesized that this PHR-based intervention would demonstrate improvements and increases, respectively in the objective and subjective domain measures. The investigators also hypothesized that engagement by study participants with MHV would be demonstrated through meeting target criteria regarding making entries into this PHR's TH function, and that participants would be satisfied with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with diagnosis of prediabetes (HbA1c 5.7-6.4%, fasting plasma glucose 100-125 mg/dL or oral glucose tolerance test 140-199 mg/dL)
* English speaking
* Access to the Internet
* Body mass index (BMI) of 25-42 kg/m and a sedentary lifestyle (not being physically active three days per week for 20 minutes each time for the previous six months and not performing regular resistance exercise)
* Able to engage in a regular program of mild-to-moderate intensity physical activity but were not currently following a weight loss diet or participating in an intervention trial

Exclusion Criteria:

* Cognitively impaired (Mini-Cog greater than or equal to 3)
* Depressed (PHQ-2 less than or equal to 3)
* Vision or hearing disorders
* Have been diagnosed with diabetes mellitus, uncontrolled hypertension, or cardiovascular disease
* Currently pregnant or nursing.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sharit, PhD, Principal Investigator — Miami VA Healthcare System, Miami, FL
Locations (1):
- Miami VA Healthcare System, Miami, FL, Miami, Florida, United States

REFERENCES:
- [Background] Sharit J, Idrees T, Andrade AD, Anam R, Karanam C, Valencia W, Florez H, Ruiz JG. Use of an online personal health record's Track Health function to promote positive lifestyle behaviors in Veterans with prediabetes. J Health Psychol. 2018 Apr;23(5):681-690. doi: 10.1177/1359105316681065. Epub 2016 Dec 5. PMID 27920356

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Health Record: The study intervention involved the provision to study participants of targeted instruction and practice on use of the Track Health function of the VA's patient health record known as My HealthyVet.
  Patient health record: The study intervention involved the provision to study participants of targeted instruction and practice on use of two features of the Track Health (TH) function of the VA's patient health record (PHR) known as My HealthyVet (MHV) -- Journals and Vitals + Readings -- for promoting positive physical activity (PA) and dietary lifestyles. Seven interactive multimedia instructional modules were developed by the study team. These modules demonstrated on a computer screen how to enter PA and diet information into the Journals feature; how to add weight data into the Vitals + Readings feature; how to view these and other measures in tabular and graphical formats over different time frames; and the concept of possible cause-effect links between behavioral lifestyle
Period: Overall Study
Arm/Group | Patient Health Record
Started | 47
Second Visit | 47 (Participants had to wear an accelerometer and make entries into their PHR over the previous 7 days.)
Completed | 38
Not Completed | 9
Not completed — Protocol Violation | 9

BASELINE CHARACTERISTICS:
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Weight
Description: measured in lbs.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: lbs.
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
lbs.
  baseline | 225.0 (36.3)
  3 months | 222.1 (36.0)
Statistical Analysis 1: Comparison: Patient Health Record; Test type: Other; p = .003, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Body Mass Index
Description: Measured in kg/m^2
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
kg/m^2
  baseline | 33.6 (3.9)
  3 months | 33.4 (3.9)

3. Primary Outcome: Change From Baseline Abdominal Circumference
Description: measured in inches
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
inches
  baseline | 44.2 (5.0)
  3 months | 43.5 (4.9)
Statistical Analysis 1: Comparison: Patient Health Record; Test type: Other; p = .007, t-test, 2 sided

4. Primary Outcome: Change From Baseline Energy Expenditure
Description: measured in kcal using an accelerometer
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
kcal
  baseline | 435.2 (208.5)
  3 months | 483.8 (221.0)
Statistical Analysis 1: Comparison: Patient Health Record; Test type: Other; p = .026, t-test, 2 sided

5. Primary Outcome: Change From Baseline Dietary Intake
Description: 24-hour dietary recall; the Nutrition Data System for Research used to compute kcal
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
kcal
  baseline | 1612.2 (598.3)
  3 months | 1525.0 (777.3)

6. Primary Outcome: Systolic and Diastolic Blood Pressure
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
mmHg
  systolic bp, baseline | 131.5 (16.6)
  systolic bp, 3 months | 124.0 (13.7)
  diastolic bp, baseline | 89.2 (10.9)
  diastolic bp, 3 moths | 81.0 (12.6)
Statistical Analysis 1: Comparison: Patient Health Record; Test type: Other; p = .003, t-test, 2 sided — systolic blood pressure
Statistical Analysis 2: Comparison: Patient Health Record; diastolic blood pressure; Test type: Other; p = .001, t-test, 2 sided

7. Secondary Outcome: Change From Baseline Physical Activity Self-efficacy
Description: an 18-item exercise self-efficacy questionnaire (confidence in one's ability to exercise) exercises); scale range: 0 - 100.
  Higher scores indicate increased self-efficacy.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
units on a scale
  baseline | 57.4 (16.8)
  3 months | 56.4 (17.5)

8. Secondary Outcome: Change From Baseline Diet Self-efficacy
Description: a single 7-point item questionnaire (confidence in one's ability to adhere to a healthy diet). Scale range: 1 - 7. Higher numbers indicate less self-efficacy.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
units on a scale
  baseline | 1.9 (1.2)
  3 months | 2.4 (1.4)
Statistical Analysis 1: Comparison: Patient Health Record; Test type: Other; p = .019, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Intent to Perform Physical Activity
Description: A single 7-point item, ranging from 1 - 7, with lower values indicating increased intent to perform physical activity
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
units on a scale
  baseline | 2.1 (1.3)
  3 months | 2.6 (1.5)

10. Secondary Outcome: Change in Intent to Adhere to Diet
Description: A single 7-point item, ranging from 1-7. Lower scores indicate an increased intent to adhere to diet
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
units on a scale
  baseline | 2.0 (1.2)
  3 months | 2.2 (1.3)

11. Secondary Outcome: Change in Patient Activation
Description: A 22-item scale that captures various domains of patient activation; scale range: 0 - 100, higher scores indicate greater activation
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Health Record
Number analyzed (Participants) | 38
units on a scale
  baseline | 67.5 (12.3)
  3 months | 67.8 (14.5)

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed.
Arm/Group | Patient Health Record
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes